CLINICAL TRIAL: NCT03202251
Title: The Impact of Deep Brain Stimulation in Patients With Lower Urinary Tract Symptoms: A Prospective, Observational, Cohort Study
Brief Title: Deep Brain Stimulation in Patients With LUTS
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Director of Research, Center for Restorative Pelvic Medicine, The Methodist Hospital Research Institute
Other Study IDs: Pro00016473
Record Dates: First submitted 2017-04-28; First posted 2017-06-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Bladder Dysfunction; Neurogenic Bladder
Keywords: overactive bladder; underactive bladder; urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Bladder, Overactive; Urinary Bladder, Underactive; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: It's is a cohort — It is a prospective, observational, cohort study

SUMMARY:
Deep brain stimulation (DBS) is a neurosurgical procedure using a device that improves motor symptoms of specific neurological and movement disorders such as Parkinson's disease or Essential Tremor. As part of the patient's care, the DBS is implanted when symptoms cannot be satisfactorily controlled with medications or conventional therapies. Lower urinary tract symptoms are common in patients who have underlying neurological or movement disorders and control over lower urinary tract function is poorly understood. In this study investigators are evaluating the effects of DBS on lower urinary tract function.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) is a neurosurgical procedure that improves motor symptoms of specific neurological and movement disorders such as Parkinson's disease or Essential Tremor. DBS is implanted when symptoms cannot be satisfactorily controlled with medications or conventional therapies. After insertion of deep electrodes, electrical stimulation will be delivered to modulate specific neurons in certain areas of the brain. Despite, the known motor effects for DBS, its nonmotor effects on other organs such as the urinary tract and bladder function remains unclear. Lower urinary tract symptoms such as frequency, urgency, urinary incontinence, or incomplete bladder emptying are common in patients who have underlying neurological or movement disorders. In addition, central neural control over lower urinary tract function is still poorly understand. In this trial investigators plan to evaluate the effects of Deep Brain Stimulators (DBS) on lower urinary tract function. This trial is designed to test the hypothesis that DBS improves objective and subjective symptoms of lower urinary tract function in specific patient populations. The investigators plan to test this hypothesis by using validated patient reported outcome questionnaires and urodynamic testing (both are part of routine care for neurogenic bladder) before and after DBS implantation. In addition, this trial will shed some light in understanding higher neural control of bladder and potentially identify target areas for future intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are a candidate for Deep Brain Stimulation (DBS) as standard care for neurologic symptoms and have a moderate or greater urinary bother American Urological Association Symptom Score (AUASS≥8)

Exclusion Criteria:

* Pregnant, breastfeeding mothers and all individuals younger than 18 years of age will be excluded. Patients with history of urinary diversion or augmentation cystoplasty will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are a candidate for therapeutic DBS because of their neurologic symptoms and have a total AUASS of ≥8.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in AUASS (American Urological Association Symptom Score) | Change in AUA symptoms score at Post DBS Implant (≥ 60 days after procedure) measurement compared to Pre-DBS (≤60 day prior to procedure) measurement.
  Subjective assessment of Deep Brain Stimulation (DBS) effect on urinary symptoms measured by AUASS questionnaire (from none= 0 to most severe=35)
Change from Baseline in I-QOL (Incontinence Quality of Life score) | Change in I-QOL score at Post DBS Implant (≥ 60 days after procedure) measurement compared to Pre-DBS (≤60 day prior to procedure) measurement.
  Subjective assessment of DBS effect on urinary incontinence related QOL measured by I-QOL questionnaire. Scores would be from 0 to 100. Higher scores indicate less impact of urinary incontinence on quality of life

SECONDARY OUTCOMES:
Change from Baseline in Neurogenic Detrusor Overactivity (NDO) | Change in Neurogenic Detrusor Overactivity pattern at Post DBS Implant (≥ 60 days after procedure) urodynamic study compared to Pre-DBS (≤60 day prior to procedure) urodynamic study.
  Using Urodynamic Study (UDS) to objectively assess DBS effect on Neurogenic Detrusor Overactivity (NDO) (Changed status from Yes to No- Yes means we see NDO at time of UDS , No means we do not see NDO at the time of UDS and we check to see if this status changes from Yes in Pre-DBS study to No in Post DBS and year 2 follow-up study ) and Bladder Compliance which is measured by diving bladder volume change to bladder pressure change (ml/cmH2O) during bladder filling at the time of UDS.
Change from baseline in Bladder Compliance | Change in bladder compliance at Post DBS Implant (≥ 60 days after procedure) urodynamic study compared to Pre-DBS (≤60 day prior to procedure) urodynamic study.
  Bladder Compliance is measured by dividing bladder volume change to bladder pressure change (ml/cmH2O) during bladder filling at the time of UDS. Bladder Compliance= ( Bladder Volume at the end of bladder filling- Bladder Volume at the beginning of bladder filling)/ Bladder Pressure at the end of bladder filling- Bladder Pressure at the beginning of bladder filling)

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined